CLINICAL TRIAL: NCT02349763
Title: Intravenous Versus Oral Regimens of Dexamethasone for Prophylaxis of Paclitaxel-associated Hypersensitivity Reaction in Primary Ovarian, Fallopian Tube and Peritoneal Cancer Patients: a Double-blind Randomized Controlled Trial
Brief Title: Dexamethasone Regimens for Prophylaxis of Paclitaxel-associated Hypersensitivity Reaction
Acronym: DEPARO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Department of Medical Services Ministry of Public Health of Thailand (Other Government)
Collaborators: Chulalongkorn University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: pHSR01
Record Dates: First submitted 2015-01-23; First posted 2015-01-29 (Estimated); Last update posted 2020-10-23 (Actual); Status verified 2015-01

CONDITIONS: Hypersensitivity Reaction
Keywords: Dexamethasone; Hypersensitivity reaction; Paclitaxel
MeSH Terms: conditions — Hypersensitivity | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Oral Dexamethasone (Active Comparator): Dexamethasone 20 mg (4 mg/tablet) or 5 tablets given orally at 12 and 6 hours before paclitaxel infusion and 0.9% NaCL (Placebo) 4 ml given intravenously at 30 minutes before paclitaxel infusion
  Interventions: Drug: Oral Dexamethasone
- Intravenous Dexamethasone (Experimental): Lactose (Placebo) 5 tablets given orally at 12 and 6 hours before paclitaxel infusion and dexamethasone 20 mg (5mg/ml) given intravenously at 30 minutes before paclitaxel infusion
  Interventions: Drug: Intravenous Dexamethasone

INTERVENTIONS:
Drug: Intravenous Dexamethasone — Lactose (Placebo) 5 tablets given orally at 12 and 6 hours before paclitaxel infusion and dexamethasone 20 mg (5mg/ml) given intravenously at 30 minutes before paclitaxel infusion
  Other Names: Dexazone
  Arms: Intravenous Dexamethasone
Drug: Oral Dexamethasone — Dexamethasone 20 mg (4 mg/tablet) or 5 tablets given orally at 12 and 6 hours before paclitaxel infusion and 0.9% NaCL (Placebo) 4 ml given intravenously at 30 minutes before paclitaxel infusion
  Other Names: Dexazone
  Arms: Oral Dexamethasone

SUMMARY:
Comparison of the efficacy and side effects of intravenous and oral regimens of dexamethasone for prophylaxis of paclitaxel-associated hypersensitivity reactions in primary ovarian, fallopian tube and peritoneal cancer patients receiving first cycle of combination paclitaxel and carboplatin.

DETAILED DESCRIPTION:
The consensus statements on the management of ovarian cancer recommended intravenous paclitaxel (175 mg/m2 over 3 hr) plus intravenous carboplatin (area under the curve [AUC] 5.0-7.5 mg/ml∙min) given every 3 weeks for six cycles for first-line chemotherapy. A major limitation of paclitaxel was its poor water solubility, which led to the use of polyoxyethylated castor oil vehicle or Cremophor® EL as diluents resulted a hypersensitivity reactions (HSRs). Initial P-HSRs generally occur within 10 minutes of the start of paclitaxel infusion and most occur with the first or second infusion. Majority of patients manifest as minor symptoms characterized by flushing and rashes but sometime life-threatening characterized by generalized urticaria, angioedema, bronchospasm and hypertension or until fatal may occur. The reaction is likely due to the release of histamine and other vasoactive substances in response to Cremophor EL. Originally, the prophylactic regimen composed of the use of an oral corticosteroid administered in two doses at 12 and 6 hours prior to paclitaxel infusion accompanied with histamine receptor H1 and H2 antagonists administered intravenously 30 minutes prior to paclitaxel infusion was found to successfully limit P-HSRs denoted as "Conventional oral prophylactic regimen".

While this three-drug prophylactic regimen has been shown to be effective, it can be inconvenient for patients because the oral corticosteroid must be taken 12 and 6 hours before chemotherapy administration. If the patient forgets to take one or both pretreatment steroid doses, it is not clear whether the patient can be safely treated. This led to the experimental prophylactic regimen of one dose of intravenous dexamethasone accompanied with the H1 and H2 antagonists administered 30 minutes prior to paclitaxel infusion was subsequently reported to be equivalent to the regimen of oral dexamethasone denoted as "Modified intravenous prophylactic regimen". This intravenous regimen results in lower total steroid doses and precludes the issues of compliance.

ELIGIBILITY:
Inclusion Criteria:

* Patient pathologically diagnosed with primary ovarian or fallopian tube or peritoneal cancer
* Patient starting a first cycle of combination paclitaxel and carboplatin at Rajavithi Hospital between February 1, 2015 and July 31, 2015
* Patient aged 18-70 years
* Patient with ECOG performance status 0-2
* Patient with the following laboratory values obtained: Hemoglobin > 10 g/dL, Absolute neutrophil count > 1500 /mm3, Platelet count > 100,000/mm3, Serum creatinine > 2.0 mg/dL, Bilirubin > 1.5 x ULN, alkaline phosphatase and SGOT > 3 x ULN
* Patient able to give free and informed consent and who agrees to participate by signing the consent form
* Patient able to speak and understand Thai
* Patient able to complete the quality of life questionnaire on Functional Assessment of Cancer Therapy - Ovarian Cancer (FACT-O) Thai version 4.0 and the personal logbook

Exclusion Criteria:

* Patient who has previously received paclitaxel or carboplatin
* Patient receiving an albumin-bound paclitaxel
* Patient who had an allergic reaction to taxanes or platinum analogues
* Patient is currently under treatment with systemic corticosteroids or has received systemic corticosteroids or histamine antagonists during the last week
* Patient who had an allergic reaction to corticosteroid or diphenhydramine or ranitidine
* Patient with severe intolerance to lactose
* Patient with an allergy or a severe intolerance to products containing castor oil e.g. cyclosporine, teniposide, diazepam, propofol

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 260 (Actual)
Dates: Start 2015-02-28 (Actual); Primary Completion 2015-07-30 (Actual); Study Completion 2015-08-30 (Actual)

PRIMARY OUTCOMES:
Incidence of Paclitaxel-Associated Hypersensitivity Reaction (P-HSRs) and severe P-HSRs (Safety endpoint) | 3 Hours after starting paclitaxel infusion
  The participants are received either intravenous dexamethasone or placebo (0.9% NaCL) at 09.30 am (30 minutes before paclitaxel infusion) depend on intervention groups. Intravenous ranitidine 50 mg and diphenhydramine 50 mg are also given all participants. Paclitaxel is started at 10.00 am by the calculated dose of is diluted in 500 ml of saline and administered by intravenous infusion over 3 hours.

SECONDARY OUTCOMES:
Incidence of side effects of dexamethasone | 1 week after completion of chemotherapy
  All participants receive the personal logbook for self-administration of side effects from dexamethasone in day 1-7
Incidence of other Adverse Events ( according to NCI CTCAE version 4.03) | Adverse events were measured at Day 1 and Day 28 of intervention
  The adverse events are collected according to NCI CTCAE version 4.03.
Quality of life (QoL) (assessed by FACT-O score) | QoL is measured at Day 0 and Day 28 of intervention
  Quality of life assessed by FACT-O score

CONTACTS AND LOCATIONS:
Overall Officials: Dr Marut Yanaranop, MD, Principal Investigator — Department of Medical Services Ministry of Public Health of Thailand
Locations (1):
- Rajavithi Hospital, Bangkok, Thailand